CLINICAL TRIAL: NCT06274099
Title: The Effect of Nursing Care Given According to Kolcaba's Comfort Theory on the Complaints and Comfort Level of Hemodialysis Patients
Brief Title: The Effect of the Care Given to Hemodialysis Patients on Comfort Level and Complaints
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reva Balci Akpinar (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Reva Balci Akpinar, Principal Investigator, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TDK-2023-12649
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis Complication; Nurse's Role
Keywords: hemodialysis; nursing care; comfort
MeSH Terms: interventions — Nursing Care

STUDY DESIGN:
Intervention Model Description: pretest posttest randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): This group will be given designated nursing care.
  Interventions: Other: nursing care
- CONTROL GROUP (Active Comparator): Routine nursing care will be provided to this group.
  Interventions: Other: nursing care

INTERVENTIONS:
Other: nursing care — It is thought that this study, in which individualized care will be based on comfort theory, will lead to individualized care in chronic diseases.

SUMMARY:
Kolcaba's comfort theory is a theory used by nurses to increase the comfort of patients. There are limited studies determining that nursing care provided according to this theory contributes to the increase in patients' comfort levels in various patient groups. This study will be carried out in the hemodialysis center of a public hospital located in the city center of Bingöl. Patients in the intervention group receiving hemodialysis treatment will be given nursing care by the researcher for 12 sessions during the sessions in which the patient receives hemodialysis treatment. In order to provide nursing care, nursing diagnoses suitable for the patient group will be determined in advance and the care the patient needs will be given according to these diagnoses.. If necessary, the researcher will add additional diagnoses to the preliminary diagnosis form and provide care.

In this research, the individual nursing care needs of the researcher patient will be determined. Individualized caregiving is unique to this study. Individually provided care is expected to increase patient comfort and satisfaction. Increased comfort will help the patient cope more easily with the disease and hemodialysis treatment symptoms. In addition, the results of individual care provided can guide nurses in their care behaviors. By adding this research to the literature, the groundwork will be laid for studies that will provide individual care to patients. It is expected that the results of this research will guide the planning of the research and the provision of individualized care in all patient groups, especially patients receiving hemodialysis treatment.

DETAILED DESCRIPTION:
American nurse theorist Katharine Kolcaba developed Comfort Theory based on the care observed or given. Kolcaba has worked in operating room, home care, and medical/surgical specialties. Kolcaba's Comfort Theory; It consists of levels of spaciousness, comfort and superiority (transcendence) and physical, psychospiritual, sociocultural and environmental dimensions. Comfort is an important goal of care that aims to provide the highest quality of life for the patient and their family. Good caregiving, family support, the way of managing information, the search for meaning in life, and the need to control life are important predictors of providing comfort. Patients' physical, sociocultural, psychospiritual and environmental problems affect their comfort. One of the treatment methods used for individuals with chronic kidney failure is Hemodialysis (HD). Living connected to a hemodialysis machine can cause physiological, psychological and social problems in sick individuals. The difficulties that patients face are that they experience physiological problems due to restriction in their nutrition, that they have to restrict fluids, that they live dependent on the treatment team, that they experience psychological problems related to changes in body image, that they experience social problems such as anxiety about the future and limitation of work life, and decreased social relations. These difficulties they experience negatively affect the daily lives and comfort of patients. Comfort is very important for patients receiving hemodialysis treatment. Nurses have important responsibilities in increasing the comfort levels and quality of life of HD patients. It is very important to plan, implement and evaluate nursing interventions .

According to Kolcaba's Comfort Theory, the results of nursing care given to children with cancer have determined that it is an appropriate approach that helps make innovative interventions to provide comfort to children with cancer and allows the patient to be evaluated holistically .

ELIGIBILITY:
Inclusion criteria:

Clinical diagnosis of chronic renal failure Receiving 3 sessions of hemodialysis treatment per week Over 18 years old Must be able to communicate

Exclusion Criteria:

Having a psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
General Comfort Scale | 4 week
  The minimum score that can be obtained from the scale is 48 and the maximum score is 192. As total score increases, comfort increases. A decrease in the score means that the comfort decreases.
Dialysis Symptom Index | 4 week
  The minimum score for the scale is 0 and the maximum score is 150. As the total score approaches 150, the effect of the symptom increases, and as it approaches 0, it indicates that the effect of the symptom decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Diğerleri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baraz S, Zarea K, Dashtbozorgi B. Comparing the effect of two educational programs on the quality of life of hemodialysis patients in iran. Iran Red Crescent Med J. 2014 Aug;16(8):e19368. doi: 10.5812/ircmj.19368. Epub 2014 Aug 5. PMID 25389489
- [Background] Borzou SR, Anosheh M, Mohammadi E, Kazemnejad A. Patients' perception of comfort facilitators during hemodialysis procedure: a qualitative study. Iran Red Crescent Med J. 2014 Jul;16(7):e19055. doi: 10.5812/ircmj.19055. Epub 2014 Jul 5. PMID 25237587
- [Background] Cabrera VJ, Hansson J, Kliger AS, Finkelstein FO. Symptom Management of the Patient with CKD: The Role of Dialysis. Clin J Am Soc Nephrol. 2017 Apr 3;12(4):687-693. doi: 10.2215/CJN.01650216. Epub 2017 Feb 1. PMID 28148557
- [Background] Ebrahimpour F, Hoseini ASS. Suggesting a Practical Theory to Oncology Nurses: Case Report of a Child in Discomfort. J Palliat Care. 2018 Oct;33(4):194-196. doi: 10.1177/0825859718763645. Epub 2018 Mar 21. PMID 29560797
- [Background] Kacaroglu Vicdan A. The Effect of Training Given to Hemodialysis Patients According to the Comfort Theory. Clin Nurse Spec. 2020 Jan/Feb;34(1):30-37. doi: 10.1097/NUR.0000000000000495. PMID 31789961
- [Background] Moledina DG, Perry Wilson F. Pharmacologic Treatment of Common Symptoms in Dialysis Patients: A Narrative Review. Semin Dial. 2015 Jul-Aug;28(4):377-83. doi: 10.1111/sdi.12378. Epub 2015 Apr 25. PMID 25913502
- [Background] Shahdadi H, Rahnama M. Experience of Nurses in Hemodialysis Care: A Phenomenological Study. J Clin Med. 2018 Feb 11;7(2):30. doi: 10.3390/jcm7020030. PMID 29439484